CLINICAL TRIAL: NCT00386633
Title: Phase I, Open, Sequential Vaccination Study on Safety and Tolerability of Two Different Doses of a Recombinant MVA HIV Polytope Vaccine (MVA-mBN32) in HIV-negative 18-50 Year Old Healthy Volunteers
Brief Title: Safety and Immunogenicity Study of Recombinant Modified Vaccinia Virus Ankara (MVA) Virus to Treat HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Monika Fluer, Bavarian Nordic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIV-POL-001
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections
Keywords: Vaccine; Safety; T-cell epitope; Acquired Immune Deficiency Syndrome Virus; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Lower dosage: 10E7_TCID50
  Interventions: Biological: MVA-mBN32
- 2 (Active Comparator): 10E8_TCID50
  Interventions: Biological: MVA-mBN32

INTERVENTIONS:
Biological: MVA-mBN32 — 3 immunizations; first study group: 10E7_TCID50
  Arms: 1
Biological: MVA-mBN32 — 3 immunizations; second study group: 10E8_TCID50
  Arms: 2

SUMMARY:
At the end of 2004 there were more than 40 million people infected worldwide with HIV, with an estimated 16,000 new infections every day (Joint United Nations Programme on HIV/AIDS [UNAIDS], 2004). The HIV epidemic threatens whole societies particularly in Africa and Asia and rates of infections in the Western countries have also increased over the last few years. However, despite more than 15 years of research, an effective vaccine against HIV and acquired immunodeficiency syndrome (AIDS) has still not been developed.

There is considerable evidence that cellular immune responses can effectively control HIV-1 replication during acute and chronic infections thereby possibly protecting individuals from infection and preventing the spread of HIV. To be truly effective in the general population, a vaccine must induce responses specific to immunologically conserved regions. The epitope-based vaccine MVA-mBN32 represents a very logical approach to this problem because of its potential to elicit a polyfunctional immune response and to focus these responses to conserved epitopes.

In this study the safety, tolerability, and immunogenicity of a recombinant MVA-BN® vaccine expressing cytotoxic T lymphocyte (CTL) and helper T lymphocyte (HTL) epitopes of HIV-1 (MVA-mBN32) in 36 healthy volunteers will be examined. This will include a full analysis of CD4+ T helper cells and CD8+ CTL responses to these epitopes, to establish the potential of such a homologous prime-boost vaccine approach to induce a broad cell-mediated response to different HIV antigens.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 50
2. Women must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to vaccination.
3. Women of childbearing potential must have used an acceptable method of contraception.
4. Troponin I within normal institutional limits.
5. Adequate renal function
6. Adequate hepatic function
7. Electrocardiogram (ECG) without abnormal findings
8. Negative HIV test for HIV-1 prior to immunization
9. HLA-A2, HLA-A3 or HLA-B7 positive.
10. Written informed consent of the subject after information of the risks and benefits of the study are provided in a language the subject clearly understands, and before any study specific procedure.
11. Ultrasound of the abdomen without clinically significant abnormalities.

Exclusion Criteria:

1. Pregnant or breast-feeding women.
2. Uncontrolled serious infection, i.e. not responding to antimicrobial therapy.
3. History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject.
4. History of or suspected or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement are not excluded.
5. Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
6. Any condition which might interfere with study objectives or would limit the subject's ability to complete the study or to be compliant in the opinion of the investigator.
7. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor.
8. History of an immediate family member (father, mother, brother, or sister) who died due to ischemic heart disease before age 50 years.
9. Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool. (http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof) NOTE: This criterion applies only to volunteers 20 years of age and older.
10. Chronic administration (defined as more than 14 days) of systemic immuno-suppressant drugs during a period starting from six months prior to administration of the vaccine and ending at study conclusion. (Corticosteroid nasal sprays are permissible. Persons who have used topical and inhaled steroids can be enrolled after their therapy is completed).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-10; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety | 40 w

CONTACTS AND LOCATIONS:
Overall Officials: Elke Jordan, PhD, Study Director — Bavarian Nordic
Locations (1):
- LMU-Munich, Department of Infectious Diseases and Tropical Medicine, Munich, Germany